CLINICAL TRIAL: NCT03160092
Title: Assessing the Feasibility of a Novel Intervention for Young People With At Risk Mental State and Attenuated Positive Psychotic Symptoms: The Viability of Its Use in the NHS and of a Future Trial
Brief Title: The Feasibility of a Novel Intervention for At Risk Mental State
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Collaborators: Norfolk and Suffolk NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212935
Record Dates: First submitted 2017-05-12; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: At Risk Mental State; Attenuated Psychotic Symptoms
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Clinical Participants will receive a 4 session individual intervention, which will be delivered by Assistant Practitioners and Assistant Psychologists (who will have received specific training in the delivering of the intervention).
  The intervention will target the participant's attenuated positive psychotic symptoms, which will be referred to as: 'unusual' experiences (unless the participant prefers an alternative).
  The therapist will focus on creating a therapeutic relationship in which the participant experiences them as warm, accepting and empathic. The aim is for the participant to feel listened to and understood.
  The intervention will focus on taking a normalising and non-catastrophising approach to the individual's unusual experiences. The participants will be provided with psychoeducation to support this aim.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — The intervention aims to:
  * Support the participant to explore their unusual experiences
  * Reduce the distress or anxiety participants feel in response to their unusual experiences, through:
    * Helping them to recognise how common these unusual experience
    * Supporting them to make sense of their unusual experiences
    * Supporting them to understand why they may be experiencing these symptoms
    * Challenging any unhelpful beliefs they hold about their symptoms
  * Help the participant to recognise the triggers to their unusual experiences
  * Support the participant to increase their activities and socialisation
  The intervention is not aiming to 'get rid' of the participant's symptoms, but to reduce their distress in response to them, which may result in improved wellbeing and reduced symptoms.

SUMMARY:
Young people with At Risk Mental State (ARMS) may have changes in their thoughts and the way they see or hear things, which they might find odd and distressing. They may be feeling tense, worried and low in mood and may not feel like socialising. They may also experience difficulties with eating and sleeping. For many people these symptoms might not last for very long, but for a small number of people, they might last longer and could become worse (health professionals call this psychosis).

Psychological therapy, which involves talking to a therapist, can help to stop these symptoms from getting worse, stopping psychosis. It can also help to make the symptoms better. Cognitive Behavioural Therapy (CBT) is the treatment that is most recommended to help young people with ARMS. But, this is not always available, can take a long time and is quite expensive. Some research has shown that brief therapy with a therapist who is warm and understanding and helps the young person to make sense of their symptoms, may be as helpful as CBT, and is quicker and cheaper.

This study hopes to develop a treatment like this and to offer it to 12 young people, aged between 16 and 25, who are experiencing the symptoms outlined. Participants will be given four treatment sessions, and will be asked to complete some questionnaires. The study aims to see how they find it and whether it seems to help them. It will also ask professionals who work with these young people what they think about the new therapy. This is a feasibility study so the findings will help us to decide whether more research should be done on this treatment and whether it could be offered in the NHS in the future.

ELIGIBILITY:
For Service User Participants (Those receiving the intervention)

Inclusion Criteria:

* 16 - 25 Years Old
* Meeting criteria for attenuated psychosis on the Comprehensive Assessment of At Risk Mental State (CAARMS; Yung et al., 2005)
* Has an allocated lead care professional within the Central Norfolk Youth Team
* Identified by their care-coordinator as having capacity and being appropriate for therapy (including not being deemed at a high risk of being a danger to themselves or others).

Exclusion Criteria:

* Meeting criteria for psychosis on the CAARMS and/or a previous open referral to an Early Intervention in Psychosis team
* Change of psychiatric medication within the previous three months
* Currently receiving psychological therapy
* Previously had Cognitive Behavioural Therapy for At Risk Mental State

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2017-11-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Assessment of At Risk Mental State (CAARMS) - Change in At Risk Symptoms | 2 months
  This is a 30 minute semi-structured interview, measuring the intensity, duration and frequency of subthreshold psychotic symptoms

SECONDARY OUTCOMES:
Clinical Outcomes in Routine Evaluation Outcome Measure (CORE-OM) - Change in psychological wellbeing | 2 months
  The CORE-OM measures: Psychological wellbeing, functioning, symptoms and risk
Revised Short Version of the Working Alliance Inventory (WAI-SR) | 2 months
  Both clinician and client versions of this measure will be used to assess the therapeutic alliance formed for each participant
Session Rating Scale (SRS) - Completed after each session | 1 week
  Used to measure the participant's views of each session

OTHER OUTCOMES:
Service User Participant Experience Questionnaire | 2 months
  Measure of the acceptability of the intervention and the study to the participants receiving the intervention (to inform the feasibility aspect of the study)
Interventional Therapist Participant Experience Questionnaire | 2 months
  Measure of the acceptability of the intervention and the study to the clinicians delivering the intervention (to inform the feasibility aspect of the study)
Youth Team Clinicians Participant Experience Questionnaire | 2 months
  Measure of the acceptability of the intervention and the study to clinicians working in NHS Youth Teams (to inform the feasibility aspect of the study)

CONTACTS AND LOCATIONS:
Locations (1):
- Central Norfolk Youth Team, 80 St Stephens Road, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No